CLINICAL TRIAL: NCT02845466
Title: Proof of Concept Study of Combined Topical Growth Factor and Protease Inhibitor in Chronic Wound Healing
Brief Title: Study of Combined Topical Growth Factor and Protease Inhibitor in Chronic Wound Healing
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: McMaster University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Lower Limb Ulcer Topical Ther
Record Dates: First submitted 2016-07-14; First posted 2016-07-27 (Estimated); Last update posted 2018-04-09 (Actual); Status verified 2018-04

CONDITIONS: Venous Ulcer; Foot Ulcer, Diabetic
Keywords: Venous Leg Ulcer; Diabetic Foot Ulcer; Wound Healing; Growth Factor; Protease Inhibitor
MeSH Terms: conditions — Varicose Ulcer; Diabetic Foot | interventions — Becaplermin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Becaplermin/Promagran Dressing (Experimental): Topical Becaplermin with a protease inhibitor wound dressing.
  Interventions: Biological: Becaplermin; Device: Promagran Dressing
- Becaplermin/Placebo Dressing (Active Comparator): Topical Becaplermin with a placebo wound dressing.
  Interventions: Biological: Becaplermin; Device: Placebo Dressing

INTERVENTIONS:
Biological: Becaplermin — 0.25 cm of 100 µg/g Becaplermin gel topically per 1cm² of ulcer area applied 3 times per week for 6 weeks.
  Other Names: Regranex
Device: Promagran Dressing — 44% oxidized regenerated cellulose (ORC), 55% collagen and 1% silver-ORC wound dressing applied 3 times per week for 4 weeks.
  Arms: Becaplermin/Promagran Dressing
Device: Placebo Dressing — Inactive wound dressing.
  Other Names: Aquacel
  Arms: Becaplermin/Placebo Dressing

SUMMARY:
Leg and foot ulcers due to venous disease or diabetes are chronic wounds that can take 6 or more months to heal. Growth factors have been used to try and improve this healing, however, many such studies have failed, and that is thought to be due enzymes in the wound that degrade the growth factors and prevent them from working. This is a proof of concept study that will evaluate the treatment of chronic leg ulcers with topically applied growth factors that are combined with a therapy to prevent their inactivation in the wound.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged ≥18 years
* Ulcer size 1-64 cm²
* Ulcer extends through both the epidermis and dermis, with no exposed tendon or bone
* Ulcer duration >3 months
* Ulcer located between and including the knee and ankle
* For venous leg ulcers - Venous refilling time <25s on photoplethysmography or abnormal venous insufficiency Duplex scan
* For diabetic foot ulcers - confirmed type 1 or type 2 diabetes mellitus with a haemoglobin A1C < 12%
* Wounds have not been treated with Promogran in the previous 4 weeks
* Patients able to give informed consent

Exclusion Criteria:

* Ankle-brachial index <0.8
* Ulcer with local or systemic signs of infection
* Patients who have been previously treated with Becaplermin gel
* Receiving corticosteroids or immune suppressants
* History of autoimmune disease
* Uncontrolled diabetes (baseline haemoglobin A1C > 12%)
* Severe rheumatoid arthritis
* Uncontrolled congestive heart failure
* Malnutrition (albumin <2.5g/dL)
* Unable to adhere to the protocol
* Known sensitivities to the wound dressings used in the trial
* A history of any previous malignancy
* pregnant or lactating women

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-08 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Level of Applied Growth Factors in Chronic Wound Fluid | 6 weeks
  The levels of the growth factors applied to the chronic wound will be measured using samples of the wound fluid gathered at the first two visits each week.

SECONDARY OUTCOMES:
Protease Levels in Chronic Wound Fluid | 6 weeks
  The levels of enzyme activity in the chronic wound will be measured using samples of the wound fluid gathered at the first two visits each week.
Chronic Wound Healing at 4 Weeks | 4 weeks
  Chronic wound healing will be measured using the VISITRAK device, which traces the outline of the chronic wound.
WOUNDCHEK Device Validity | 6 weeks
  The WOUNDCHEK device will be used in order to test for levels of enzyme activity in the chronic wound. This data will then be compared to the enzyme activity as determined by the levels analyzed in the chronic wound fluid.
Levels of Healing Biomarkers in Chronic Wound Fluid | 6 weeks
  The levels of the potential biomarker of healing GMCSF in the chronic wound fluid will be measured using samples of the chronic wound fluid collected at the first two visits each week.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Stacey, MBBS, Doctor of Surgery, Principal Investigator — McMaster University
Locations (1):
- Hamilton General Hospital, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stacey M. Combined Topical Growth Factor and Protease Inhibitor in Chronic Wound Healing: Protocol for a Randomized Controlled Proof-of-Concept Study. JMIR Res Protoc. 2018 Apr 27;7(4):e97. doi: 10.2196/resprot.8327. PMID 29703712